CLINICAL TRIAL: NCT06876467
Title: Etude de la réponse Cellulaire Induite Post-vaccination Contre le Virus de l'hépatite B
Brief Title: Study of the Cellular Response Induced After Vaccination Against the Hepatitis B Virus
Acronym: HBVax
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APH241703
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis B Vaccination; Immune Response; T Cells
Keywords: PBMCs isolation; Serology; Spectral cytometry; RNA sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals receiving HBV vaccination
  Interventions: Other: Evaluation of cellular response

INTERVENTIONS:
Other: Evaluation of cellular response — detection of HBsAg-specific T lymphocytes by spectral cytometry

SUMMARY:
296 million people worldwide are infected with the hepatitis B virus (HBV), despite the existence of an effective prophylactic vaccine. Current treatments (nucleoside analogues and pegylated interferon-α) do not prevent chronic hepatitis B (CHB) patients from developing liver fibrosis or hepatocellular carcinoma.

Vaccination is the best way to prevent HBV infection. The first generation of plasma-based vaccines, introduced in the 1980s, has now been superseded by protein vaccines, which are the only ones authorized in France. They are safe and effective. After an initial series of three out of four doses, protective levels of antibodies to the HBV surface antigen (anti-HBsAg; ≥10 IU/mL) are achieved in over 95% of infants, children and young adults.

HBV antigen (Ag)-specific CD4+ and CD8+ T lymphocytes play a major role in the control of HBV infection, contributing to viral clearance and the pathophysiology of acute hepatitis B. However, during HBC, these HBV-specific T cells develop a dysfunctional phenotype and become 'exhausted'. T lymphocytes directed against surface protein antigens (HBsAg) are the most affected by depletion mechanisms - these disappear completely in chronically infected patients, suggesting an important role for these T lymphocytes in infection control. Interestingly, recent studies of rare patients undergoing functional recovery from chronic infection following antiviral treatment have shown a re-emergence of T lymphocytes directed against HBsAg, confirming the importance of these cells in controlling viral replication. Although the protection induced by hepatitis B vaccination has mainly been attributed to the humoral response, a few studies have documented the presence of HBsAg-specific T lymphocytes. These could contribute to the maintenance of a long-term post-vaccination humoral response. The aim of this study is therefore to determine the frequency of healthy individuals receiving HBV vaccination who have a detectable HBsAg-specific T-cell response post-vaccination. We will also study the potential correlation between the frequency of HBsAg-specific T lymphocytes and the level of serum anti-HBsAg antibodies, and we will finely characterize the functional phenotype of these cells using cutting-edge methods and technologies (spectral cytometry, sequencing of mRNA and TCRs). These data will contribute to a better understanding of the biological mechanisms associated with HBV vaccine-induced protection.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Pre-vaccination HBV serology carried out within 4 weeks prior to vaccination
* Collection of no objection

Exclusion Criteria:

* Opposition of the person or inability to give opposition
* Pregnant or breast-feeding women
* Chronic illnesses affecting the individual's immune system (asplenia; hyposplenia; haematological cancer; auto-immune disease requiring immunosuppressive treatment, HIV infection).
* Non-affiliation with a social security scheme, Universal Medical Coverage or any equivalent scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals receiving HBV vaccination
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with a cellular response | At inclusion
  Proportion of individuals with a cellular response directed against HBsAg following HBV vaccination At inclusion, 5 to 10 weeks after HBV vaccination

SECONDARY OUTCOMES:
Frequency of pehotypes of T lymphocytes post-HBV vaccination | At inclusion
  Phenotypic and functional characterization of HBsAg-specific CD4+ and CD8+ T lymphocytes post-HBV vaccination Quantitative results obtained by spectral cytometry and RNA sequencing to characterise HBsAg-specific LTs 5 to 10 weeks after HBV vaccination
Anti-HBsAg antibody levels | At inclusion
  Before and after vaccination 4 weeks prior to vaccination and 5 to 10 weeks after vaccination
Percentage of LT CD4 circulating cells | At inclusion
  5 to 10 weeks after vaccination
Percentage of LT CD8 circulating cells | At inclusion
  5 to 10 weeks after vaccination

IPD SHARING:
Plan to Share IPD: Undecided